CLINICAL TRIAL: NCT01887600
Title: A Phase 3, Randomized, Double-Blind, Placebo Controlled Study of the Efficacy and Safety of Roxadustat for the Treatment of Anemia in Chronic Kidney Disease Patients Not on Dialysis
Brief Title: Roxadustat in the Treatment of Anemia in Chronic Kidney Disease Patients Not Requiring Dialysis
Acronym: ALPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Collaborators: Kyntra Bio (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1517-CL-0608; 2012-005180-27 (EudraCT Number)
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-10

CONDITIONS: Anemia in Chronic Kidney Disease in Non-dialysis Patients
Keywords: anemia; chronic kidney disease (CKD); Hemoglobin (Hb); non-dialysis
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — roxadustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Roxadustat (Experimental): Participants received roxadustat according to the tiered weight-based approach, with starting doses of 70 mg given thrice weekly (TIW) to participants weighing up to 70 kg and 100 mg given TIW to participants weighing more than 70 kg. Dose-titration was performed based upon regular measurement of Hb levels until participants achieved central Hb value of ≥ 11.0 g/dL and Hb increase from baseline (BL) of ≥ 1.0 g/dL at two consecutive study visits, separated by at least 5 days. Once target Hb level was reached participants entered maintenance period during which roxadustat dosage was adjusted every 4 weeks to maintain participants Hb level within the target range of 10.0 g/dL and 12.0 g/dL. Participants received roxadustat for at least 52 weeks up to a maximum of 104 weeks.
  Interventions: Drug: Roxadustat
- Placebo (Placebo Comparator): Participants received matching placebo according to the tiered weight-based approach, with starting doses of 70 mg given thrice weekly (TIW) to participants weighing up to 70 kg and 100 mg given TIW to participants weighing more than 70 kg. Dose-titration was performed based upon regular measurement of Hb levels until participants achieved central Hb value of ≥ 11.0 g/dL and Hb increase from baseline (BL) of ≥ 1.0 g/dL at two consecutive study visits, separated by at least 5 days. Once target Hb level was reached participants entered maintenance period during which roxadustat dosage was adjusted every 4 weeks to maintain participants Hb level within the target range of 10.0 g/dL and 12.0 g/dL. Participants received matching placebo for at least 52 weeks up to a maximum of 104 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roxadustat — Roxadustat was administered initially according to the tiered weight-based dosing, where participants with weight from ≥ 45 to ≤ 70 kg received 70 mg and participants with > 70 to ≤ 160 kg received 100 mg of roxadustat. Dose-titration based upon regular measurement of Hb levels was performed until participants achieved central Hb value of ≥ 11.0 g/dL and Hb increase from baseline (BL) of ≥ 1.0 g/dL at two consecutive study visits, separated by at least 5 days. Once target Hb level was reached participants entered maintenance period during which roxadustat dosage was adjusted every 4 weeks to maintain participants Hb level within the target range of 10.0 g/dL and 12.0 g/dL.
  Other Names: ASP1517; FG-4592
  Arms: Roxadustat
Drug: Placebo — Placebo was administered initially according to the tiered weight-based dosing, where participants with weight from ≥ 45 to ≤ 70 kg received 70 mg and participants with > 70 to ≤ 160 kg received 100 mg of roxadustat. Dose-titration based upon regular measurement of Hb levels was performed until participants achieved central Hb value of ≥ 11.0 g/dL and Hb increase from baseline (BL) of ≥ 1.0 g/dL at two consecutive study visits, separated by at least 5 days. Once target Hb level was reached participants entered maintenance period during which roxadustat dosage was adjusted every 4 weeks to maintain participants Hb level within the target range of 10.0 g/dL and 12.0 g/dL.
  Arms: Placebo

SUMMARY:
This study was conducted to treat anemia in patients with chronic kidney disease. Anemia is a reduced number of red blood cells or hemoglobin. Hemoglobin is important for the transport of oxygen in your blood. The purpose of the study was to see if Roxadustat is both effective and safe as a treatment for anemia in patients with chronic kidney disease.

DETAILED DESCRIPTION:
The study consisted of three study periods as follows:

* Screening period: up to 6 weeks
* Treatment period: minimum 52 weeks (primary treatment period) up to a maximum of 104 weeks (extended treatment period)
* Post-Treatment Follow-Up period: 4 weeks

ELIGIBILITY:
Inclusion criteria:

* Participant has a diagnosis of chronic kidney disease, with Kidney Disease Outcomes Quality Initiative (KDOQI) Stage 3, 4 or 5, not receiving dialysis; with an Estimated Glomerular Filtration Rate (eGFR) <60 mL/min/1.73 m^2 estimated using the abbreviated 4-variable Modification of Diet in Renal Disease (MDRD) equation.
* The mean of the Participant's three most recent Hb values during the Screening period, obtained at least 4 days apart, must be less than or equal to 10.0 g/dL, with a difference of less than or equal to 1.0 g/dL between the highest and the lowest values. The last Hb value must be within 10 days prior to randomization.
* Participant has a ferritin level greater than or equal to 30 ng/mL (greater than or equal to 67.4 pmol/L) at screening.
* Participant has a transferrin saturation (TSAT) level greater than or equal to 5% at screening.
* Participant has a serum folate level greater than or equal to lower limit of normal at screening.
* Participant has a serum vitamin B12 level greater than or equal to lower limit of normal at screening.
* Participant's alanine aminotransferase (ALT), aspartate aminotransferase (AST) levels are less than or equal to 3 x upper limit of normal (ULN), and total bilirubin (TBL) is less than or equal to 1.5 x ULN.
* Participant's body weight is 45.0 kg up to a maximum of 160.0 kg.

Exclusion criteria:

* Participant has received any ESA treatment within 12 weeks prior to randomization.
* Participant has had more than one dose of IV iron within 12 weeks prior to randomization.
* Participant has received a RBC transfusion within 8 weeks prior to randomization.
* Participant has a known history of myelodysplastic syndrome or multiple myeloma.
* Participant has a known hereditary hematologic disease such as thalassemia or sickle cell anemia, pure red cell aplasia, or other known causes for anemia other than CKD.
* Participant has a known hemosiderosis, hemochromatosis, coagulation disorder, or hypercoagulable condition.
* Participant has chronic inflammatory disease that could impact erythropoiesis (e.g., systemic lupus erythematosus, rheumatoid arthritis, celiac disease) even if it is currently in remission.
* Participant is anticipated to have elective surgery that is expected to lead to significant blood loss or anticipated elective coronary revascularization.
* Participant has active or chronic gastrointestinal bleeding.
* Participant has received any prior treatment with roxadustat or a hypoxia-inducible factor Prolyl Hydroxylase Inhibitor (HIF-PHI).
* Participant has been treated with iron-chelating agents within 4 weeks prior to randomization.
* Participant has a history of chronic liver disease (e.g., cirrhosis or fibrosis of the liver)
* Participant has a known New York Heart Association Class III or Intravenous (IV) congestive heart failure.
* Participant has had a myocardial infarction, acute coronary syndrome, stroke, seizure, or a thrombotic/thromboembolic event (e.g., pulmonary embolism) within 12 weeks prior to randomization.
* Uncontrolled hypertension or two or more blood pressure (BP) values of systolic BP (SBP) greater than or equal to 160 mmHg or diastolic BP (DBP) greater than or equal to 95 mmHg confirmed by repeat measurement within 2 weeks prior to randomization.
* Participant has a diagnosis or suspicion (e.g., complex kidney cyst of Bosniak Category 2F or higher) of renal cell carcinoma on renal ultrasound within 12 weeks prior to randomization.
* Participant has a history of malignancy, except the following: cancers determined to be cured or in remission for greater than or equal to 5 years, curatively resected basal cell or squamous cell skin cancers, cervical cancer in situ, or resected colonic polyps.
* Participant is positive for any of the following: Human Immunodeficiency Virus (HIV); hepatitis B surface antigen (HBsAg); or anti-hepatitis C virus antibody (anti-HCV Ab).
* Participant has an active clinically significant infection manifested by White Blood Count (WBC) > ULN, and/or fever, in conjunction with clinical signs or symptoms of infection within one week prior to randomization.
* Participant has a known untreated proliferative diabetic retinopathy, diabetic macular edema, macular degeneration and retinal vein occlusion.
* Participant has had any prior organ transplant (that has not been explanted) or a scheduled organ transplantation.
* Participant has participated in any interventional clinical study or has been treated with any investigational drugs within 30 days or 5 half lives or limit set by national law, whichever is longer, prior to the initiation of Screening.
* Participant has an anticipated use of dapsone in any dose amount or chronic use of acetaminophen (paracetamol) > 2.0 g/day during the treatment or follow-up period of the study.
* Participant has a history of alcohol or drug abuse within 2 years prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Actual)
Dates: Start 2013-09-03 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Chair — Astellas Pharma Europe B.V.
Locations (138):
- Belarus (7):
  - Site BY37503, Brest
  - Site BY37501, Grodno
  - Site BY37504, Homyel
  - Site BY37506, Minsk
  - Site BY37507, Minsk
  - Site BY37505, Minsk
  - Site BY37502, Vitebsk
- Belgium (6):
  - Site BE32004, Brussels, Flemish Brabant
  - Site BE32002, Antwerp
  - Site BE32012, Baudour
  - Site BE32017, Bonheiden
  - Site BE32014, Ieper
  - Site BE32013, Liège
- Bulgaria (7):
  - Site BG35923, Pazardzhik
  - Site BG35906, Sofia
  - Site BG35908, Sofia
  - Site BG35910, Sofia
  - Site BG35907, Stara Zagora
  - Site BG35916, Varna
  - Site BG35903, Veliko Tarnovo
- Colombia (3):
  - Site CO57007, Barranquilla
  - Site CO57008, Barranquilla
  - Site CO57002, Pereira
- Dominican Republic (4):
  - Site DO17101, La Fe Santo Domingo
  - Site DO17102, Santiago de los Caballeros
  - Site DO17104, Santo Domingo
  - Site DO17103, Santo Domingo
- Site EE37201, Tallinn, Estonia
- Georgia (3):
  - Site GE99503, Tbilisi
  - Site GE99504, Tbilisi
  - Site GE99502, Tbilisi
- Greece (3):
  - Site GR30003, Heraklion
  - Site GR30002, Pátrai
  - Site GR30001, Thessaloniki
- Guatemala (8):
  - Site GT50209, Chiquimula
  - Site GT50205, Guatemala City
  - Site GT50206, Guatemala City
  - Site GT50203, Guatemala City
  - Site GT50202, Guatemala City
  - Site GT50208, Guatemala City
  - Site GT50207, Guatemala City
  - Site GT50201, Guatemala City
- Hungary (7):
  - Site HU36029, Budapest
  - Site HU36025, Győr
  - Site HU36026, Kaposvár
  - Site HU36027, Kistarcsa
  - Site HU36008, Pécs
  - Site HU36028, Szent
  - Site HU36003, Zalsaegerszeg
- Italy (5):
  - Site IT39001, Bari
  - Site IT39008, Lecco
  - Site IT39006, Milan
  - Site IT39037, Modena
  - Site IT39036, Pavia
- Panama (2):
  - Site PA50703, Colón
  - Site PA50701, Panama City
- Peru (2):
  - Site PE51001, Iquitos
  - Site PE51002, Trujillo
- Poland (11):
  - Site PL48001, Krakow, Malopolska
  - Site PL48002, Katowice
  - Site PL48012, Lodz
  - Site PL48008, Lodz
  - Site PL48057, Nowy Tomyśl
  - Site PL48013, Szczecin
  - Site PL48007, Tarnów
  - Site PL48005, Warsaw
  - Site PL48004, Warsaw
  - Site PL48006, Wroclaw
  - Site PL48014, Zamość
- Romania (6):
  - Site RO40005, Timișoara, Timiș County
  - Site RO40001, Brasov
  - Site RO40021, Bucharest
  - Site RO40012, Bucharest
  - Site RO40003, Bucharest
  - Site RO40004, Oradea
- Russia (20):
  - Site RU70024, Chelyabinsk
  - Site RU70054, Irkutsk
  - Site RU70008, Kaluga
  - Site RU70051, Moscow
  - Site RU70007, Moscow
  - Site RU70005, Moscow
  - Site RU70048, Moscow
  - Site RU70047, Moscow
  - Site RU70003, Nizhny Novgorod
  - Site RU70004, Omsk
  - Site RU70043, Petrozavodsk
  - Site RU70014, Rostov-on-Don
  - Site RU70022, Saint Petersburg
  - Site RU70045, Saint Petersburg
  - Site RU70011, Saint Petersburg
  - Site RU70002, Saint Petersburg
  - Site RU70060, Saratov
  - Site RU70006, Smolensk
  - Site RU70057, Yaroslavl
  - Site RU70001, Yaroslavl
- Serbia (7):
  - Site RS38102, Belgrade
  - Site RS38104, Belgrade
  - Site RS38105, Belgrade
  - Site RS38103, Belgrade
  - Site RS38117, Kruševac
  - Site RS38101, Niš
  - Site RS38116, Zrenjanin
- South Africa (6):
  - Site ZA27001, Observatory, Cape Town
  - Site ZA27004, Bloemfontein, Free State
  - Site ZA27002, Durban, KwaZulu-Natal
  - Site ZA27008, Durban
  - Site ZA27006, Parow
  - Site ZA27007, Port Elizabeth
- Spain (6):
  - Site ES34010, Alcorcón, Madrid
  - Site ES34011, Galdakao, Vizcaya
  - Site ES34002, Badalona-Barcelona
  - Site ES34003, Barcelona
  - Site ES34006, Barcelona
  - Site ES34007, Ciudad Real
- Turkey (Türkiye) (4):
  - Site TR90003, Ankara
  - Site TR90016, Edirne
  - Site TR90024, Kocaeli
  - Site TR90020, Malatya
- Ukraine (16):
  - Site UA38009, Lviv, Lvivska
  - Site UA38021, Cherkasy
  - Site UA38003, Chernivtsi
  - Site UA38006, Dnipro
  - Site UA38016, Ivano-Frankivsk
  - Site UA38011, Kharkiv
  - Site UA38015, Kherson
  - Site UA38010, Kyiv
  - Site UA38012, Kyiv
  - Site UA38017, Kyiv
  - Site UA38007, Mykolaiv
  - Site UA38008, Odesa
  - Site UA38019, Odesa
  - Site UA38001, Ternopil
  - Site UA38018, Uzhhorod
  - Site UA38002, Zaporizhzhya
- United Kingdom (4):
  - Site GB44008, Cambridge
  - Site GB44001, Swansea
  - Site GB44005, Welwyn Garden City
  - Site GB44004, Westcliff-on-Sea

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Provenzano R, Szczech L, Leong R, Saikali KG, Zhong M, Lee TT, Little DJ, Houser MT, Frison L, Houghton J, Neff TB. Efficacy and Cardiovascular Safety of Roxadustat for Treatment of Anemia in Patients with Non-Dialysis-Dependent CKD: Pooled Results of Three Randomized Clinical Trials. Clin J Am Soc Nephrol. 2021 Aug;16(8):1190-1200. doi: 10.2215/CJN.16191020. PMID 34362786
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=363

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study population consisted of anemic participants with stages 3, 4 or 5 chronic kidney disease (CKD) (Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m^2) who were not on dialysis. Participants were recruited from 125 study centers located in 22 countries.
Pre-assignment Details: A total of 594 participants with CKD were randomized to one of the 2 treatment arms in a 2:1 ratio receiving roxadustat or placebo. Anemia was defined as a mean Hb ≤ 10.0 g/dL upon repeated measurements during the screening period. Participants needed a ferritin ≥30 ng/mL (≥ 67.4 pmol/L) and transferrin saturation (TSAT) ≥ 5%.
Period: Overall Study
Arm/Group | Roxadustat | Placebo
Started | 391 | 203
Treatment Received | 391 | 203
Completed | 245 | 89
Not Completed | 146 | 114
Not completed — Death | 39 | 16
Not completed — Lack of Efficacy | 3 | 26
Not completed — Lost to Follow-up | 5 | 1
Not completed — Physician Decision | 7 | 8
Not completed — Protocol Deviation | 3 | 0
Not completed — Withdrawal by Subject | 58 | 52
Not completed — Adverse Event | 21 | 9
Not completed — Non-compliance with study drug | 3 | 0
Not completed — Miscellaneous | 6 | 2
Not completed — Progressive Disease | 1 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population was the All Randomized, which consisted of participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Roxadustat | Placebo | Total
Number analyzed (Participants) | 391 | 203 | 594
Age, Continuous [Mean (Standard Deviation); unit: Year] | 60.6 (13.5) | 61.7 (13.8) | 61.0 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 222 | 104 | 326
  Male | 169 | 99 | 268
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 0 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 3 | 13
  White | 335 | 182 | 517
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 37 | 18 | 55
History of Diabetes (Type 1 or 2) [Count of Participants; unit: Participants]
  Yes | 146 | 89 | 235
  No | 245 | 114 | 359
Iron Repletion at Baseline [Count of Participants; unit: Participants]
  TSAT >= 20% and Ferritin >= 100 ng/mL | 204 | 109 | 313
  TSAT < 20% or Ferritin < 100 ng/mL | 187 | 94 | 281
Baseline Hemoglobin (Hb) Value [Mean (Standard Deviation); unit: g/dL] — Baseline Hb was defined as the mean of four latest central laboratory Hb values prior or on the same date as first study drug intake (pre-dose).
  g/dL | 9.08 (0.76) | 9.10 (0.72) | 9.08 (0.75)
Baseline Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] — eGFR was derived using the modification of diet in renal disease formula (MDRD).
  mL/min/1.73m^2 | 16.5 (10.2) | 17.2 (11.7) | 16.7 (10.7)
Time From Chronic Kidney Disease (CKD) Diagnosis [Mean (Standard Deviation); unit: Years] | 5.65 (7.02) | 4.91 (5.99) | 5.40 (6.69)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Hemoglobin (Hb) Response to Treatment at Two Consecutive Visits During the First 24 Weeks of Treatment Without Rescue Therapy Prior to Hb Response
Description: Hemoglobin (Hb) response was measured as Yes or No. Response Yes (responders) was defined as: Hb ≥11.0 g/dL and Hb increase from baseline by ≥ 1.0 g/dL, for participants with baseline Hb > 8.0 g/dL; or Hb increase from baseline by ≥ 2.0 g/dL, for participants with baseline Hb ≤ 8.0 g/dL at two consecutive visits with available data separated at least 5 days during the first 24 weeks of treatment without having received rescue therapy (red blood cell (RBC) transfusion, erythropoiesis-stimulating agent (ESA), or intravenous (IV) iron prior to Hb response. This was the primary efficacy endpoint for EU (EMA).
Time Frame: Baseline to week 24
Population: The analysis population was the full analysis set (FAS), which consisted of all randomized participants who received at least one dose of study drug and had at least one post-dose Hb assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
Percentage of Participants | 79.2 [74.8 to 83.1] | 9.9 [6.1 to 14.8]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; The Cochran-Mantel-Haenszel (CMH) test was adjusted by region, history of of cardiovascular, cerebrovascular or thromboembolic (CV) disease, baseline Hb and baseline estimated glomerular filtration rate (eGFR). Superiority of roxadustat versus placebo was to be declared if the lower bound of the two-sided 95% confidence interval of the CMH odds ratio was higher than 1; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 34.74, 95% CI 2-sided [20.48 to 58.93] — Please note Odds Ratio and CI are shown in percentages

2. Primary Outcome: Hb Change From Baseline (BL) to the Average Hb in Weeks 28-52 Regardless of Rescue Therapy
Description: The change from baseline to the average Hb values across weeks 28 to 52 without having received rescue therapy. The Hb values from visit windows at weeks 28, 32, 36, 40, 44, 48 and 52 were used for the calculation of the average of weeks 28 to 52. This was the primary efficacy endpoint for US (FDA).
Time Frame: Baseline and weeks 28 to 52
Population: The analysis population was All Randomized, and it consisted of all randomized participants with available data at all time points.
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 312 | 146
g/dL | 1.992 [1.82 to 2.16] | 0.300 [0.09 to 0.51]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; The Analysis of Covariance (ANCOVA) with Multiple Imputations (MI) model, adjusting for covariates was used for the analysis. The model included treatment as fixed factor, region and history of CV disease as class factors and baseline Hb, baseline eGFR as continuous covariates. Superiority of roxadustat versus placebo was considered successful if the lower bound of the two-sided 95% confidence interval of the difference between treatment arms (roxadustat minus placebo) was higher than 0; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = 1.692, 95% CI [1.52 to 1.86]

3. Secondary Outcome: Hb Change From BL to the Average Hb in Weeks 28-36 Without Having Received Rescue Therapy Within 6 Weeks Prior to and During 8-Week Evaluation Period
Description: The Hb values from visit windows at weeks 28, 32 and 36 were used for the calculation of the average of weeks 28 to 36.
Time Frame: Baseline and weeks 28 to 36
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 311 | 139
g/dL | 2.069 [1.94 to 2.20] | 0.470 [0.30 to 0.64]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; The model includes treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit interaction as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences. Tested using a fixed sequence testing procedure to maintain the overall two-sided type I error rate at 0.05; Least squares mean difference = 1.599, 95% CI 2-sided [1.41 to 1.78]

4. Secondary Outcome: Change From BL in Low-Density Lipoprotein (LDL) Cholesterol (Regardless of Fasting Status) to the Average LDL Cholesterol of Weeks 12 to 28
Description: Analysis was completed on all values collected on day 1 and weeks 12, 20 and 28.
Time Frame: Baseline and weeks 12 to 28
Population: The analysis population was the FAS, which consisted of all randomized participants who received at least one dose of study drug and had at least one post-dose Hb assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 342 | 185
mmol/L | -0.650 [-0.76 to -0.54] | 0.051 [-0.08 to 0.18]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; A Mixed Model of Repeated Measures has been applied up to week 28. The results were based on the estimated difference between the two treatment arms and overall mean effects during the period (weeks 12 to 28). The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb, baseline eGFR and baseline LDL as continuous variables; Test type: Superiority — Superiority of roxadustat versus placebo was considered successful if the upper bound of the two-sided 95% confidence interval of the difference between treatment arms (roxadustat minus placebo) is below 0; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Least squares mean difference = -0.701, 95% CI [-0.83 to -0.57]

5. Secondary Outcome: Time to First Use of Rescue Therapy (Composite of Red Blood Cell (RBC) Transfusions, Erythropoiesis-stimulating Agent (ESA) Use, and Intravenous (IV) Iron)
Description: The time to first use of rescue therapy was calculated (in years) as: (First event date - Analysis date of first dose intake + 1) / 365.25. The First event date was defined as Date of first dose of rescue medication during the efficacy emergent period and Analysis date of first dose intake was defined as date of first study drug dose intake collected on day 1. The Efficacy Emergent Period was defined as the evaluation period from the analysis date of first dose intake up to 7 days after the analysis date of last dose or the end of treatment (EOT) visit, whichever occurred first. Data reported was analysed by Kaplan-Meier estimate for cumulative proportion. Medication onset date was the date of the first use of rescue medication.
Time Frame: Baseline to week 104 (End of Treatment [EOT])
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
Percentage of participants
  Year 0.5 | 6.1 [3.6 to 8.7] | 33.3 [26.5 to 40.1]
  Year 1 | 13.0 [9.3 to 16.7] | 50.1 [42.4 to 57.7]
  Year 1.5 | 22.0 [16.6 to 27.3] | 52.5 [44.5 to 60.5]
  Year 2 | 26.3 [20.2 to 32.4] | 57.8 [48.7 to 66.9]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Hazard ratio was calculated using stratified Cox Proportional Hazards Regression stratifying on CV history and region and adjusting on Hb and eGFR at baseline as continuous covariates. Superiority is declared if the upper bound of the 95% CI is below 1.0; Test type: Superiority; p < 0.001, Regression, Cox — Tested using a fixed sequence testing procedure to maintain the overall two-sided type I error rate at 0.05; Hazard Ratio (HR) = 0.238, 95% CI 2-sided [0.17 to 0.33]

6. Secondary Outcome: Change From BL in Short Form (SF)-36 Vitality (VT) Sub-score to the Average VT Sub-score of Weeks 12 to 28
Description: Change from BL in SF-36 VT sub-score to the average value in weeks 12-28 was calculated using the physical component scores (PCS) of SF-36. The multi-purpose, short-form health survey has 36 questions with an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures. The survey measures eight dimensions or scales: (1) physical functioning (PF) (10 items); (2) role limitations due to physical health problems (RP) (3 items); (3) bodily pain (BP) (2 items); (4) social functioning (SF) (2 items); (5) general health perceptions (GH) (5 items); (6) role limitations due to emotional problems (RE) (3 items); (7) vitality, energy or fatigue (VT) (4 items); and (8) mental health (MH) (5 items). The SF-36 scores ranged from 0-100 with higher scores indicating better health status.
Time Frame: Baseline and weeks 12 to 28
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 340 | 185
Units on a Scale | 2.788 [1.56 to 4.01] | 1.661 [0.23 to 3.10]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; A Mixed Model of Repeated Measures has been applied using the visits up to week 28. The results were based on the estimated difference between the two treatment arms and overall mean effects throughout the evaluation period (weeks 12 to 28). The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline SF-36 VT, baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p = 0.093, Mixed Models Analysis — LSM Difference p-value is for test of differences.Tested using a fixed sequence testing procedure to maintain the overall two-sided type I error rate at 0.05; Least squares mean difference = 1.127, 95% CI 2-sided [-0.19 to 2.44]

7. Secondary Outcome: Change From BL in SF-36 Physical Functioning (PF) Sub-score to the Average PF Sub-score of Weeks 12 to 28
Description: Change from baseline in SF-36 PF normalized sub-score compared to the average PF sub-score of weeks 12 to 28. The multi-purpose, short-form health survey has 36 questions with an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures. Change from baseline in PF sub score of SF-36 to the average of weeks 12-28 was compared by treatment arm for all participants (primary analysis) and in the subsets of participants with baseline PF sub score below 35 and equal or above 35. The SF-36 scores ranged from 0-100 with higher scores indicating better health status. All available SF-36 PF values were used i.e., both scheduled and unscheduled for the calculation of the average PF sub-score of weeks 12 to 28.
Time Frame: Baseline and weeks 12 to 28
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 340 | 185
Units on a Scale | 1.344 [0.15 to 2.54] | 0.632 [-0.76 to 2.03]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; A Mixed Model of Repeated Measures has been applied using the visits up to week 28. The results were based on the estimated difference between the two treatment arms and overall mean effects throughout the evaluation period (weeks 12 to 28). The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline SF-36 PF, baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p = 0.27, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Least squares mean difference = 0.713, 95% CI 2-sided [-0.56 to 1.98]

8. Secondary Outcome: Change From BL in Mean Arterial Pressure (MAP) to the Average MAP of Weeks 20 to 28
Description: The MAP was derived for each visit from the average systolic (SBP) and diastolic blood pressure (DBP) calculated for each visit using the three readings and the following equation: MAP = (2/3) * DBP + (1/3) * SBP. Baseline assessment was the assessment on day 1 (average of the three readings). If the baseline assessment was missing, then the latest available value prior to first drug administration was used.
Time Frame: Baseline and weeks 20 to 28
Population: The analysis population was the per protocol set (PPS), which consisted of all FAS participants who did not meet any reasons for exclusion from the PPS and had all available data at all time points.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 310 | 146
mmHg | -0.814 [-1.83 to 0.20] | -1.656 [-2.91 to -0.41]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Mixed Model of Repeated Measures was applied using the visits up to week 28. The results were based on the estimated difference between the two treatment arms with overall mean effects throughout the evaluation period (weeks 20 to 28). The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline MAP, baseline Hb, baseline eGFR as continuous covariates; Test type: Non-Inferiority — Non-inferiority can be concluded if the upper bound of the two-sided 95% CI of the difference between roxadustat and placebo (roxadustat minus placebo) is below 2 mmHg; p = 0.182, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 0.842, 95% CI 2-sided [-0.40 to 2.08]

9. Secondary Outcome: Time to First Occurrence of Hypertension
Description: Occurrence of hypertension was defined as SBP increase from BL ≥20 mmHg and SBP >170 mmHg or DBP increase from BL ≥15 mmHg and DBP ≥110 mmHg. Time to first occurrence of hypertension was defined as first date where SBP criterion or DBP criterion is met, whichever occurred first. Data was analysed using Kaplan-Meier estimate for cumulative proportion.
Time Frame: Baseline and year 0.5, year 1, year 1.5 and year 2
Population: The analysis population was the PPS, which consisted of all FAS participants who did not meet any reasons for exclusion from the PPS and had all available data at all time points.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 359 | 183
Percentage of participants
  Year 0.5 | 11.4 [7.9 to 14.8] | 10.1 [5.5 to 14.7]
  Year 1 | 14.8 [10.9 to 18.8] | 12.5 [7.3 to 17.7]
  Year 1.5 | 17.5 [13.0 to 21.9] | 12.5 [7.3 to 17.7]
  Year 2 | 18.5 [13.7 to 23.3] | 12.5 [7.3 to 17.7]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Hazard ratio was calculated using stratified Cox Proportional Hazards Regression stratifying on CV history and region and adjusting on Hb and eGFR at baseline as continuous covariates; Test type: Non-Inferiority — Non-inferiority is declared if the upper bound of the 95% CI is below 1.3 (hazard ratio); p = 0.334, Regression, Cox; Hazard Ratio (HR) = 1.290, 95% CI 2-sided [0.77 to 2.16]

10. Secondary Outcome: Rate of Progression of CKD Measured by Annualized Estimated Glomerular Filtration Rate (eGFR) Slope Over Time
Description: Annualized eGFR slope over time was estimated by a random slopes and intercepts model using all available eGFR values (one baseline and all post-treatment values up to EOT period or start of dialysis adjusted on baseline Hb, region, CV history at baseline and the interaction terms (baseline eGFR by timepoint and baseline Hb by timepoint). All assessments collected after initiation of chronic dialysis (acute or chronic) are excluded from the analysis. Baseline assessment was the assessment from day 1 visit. If this value was missing, the value from screening visit was used.
Time Frame: Baseline to week 108
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: ml/min per 1.73 m^2 per year
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
ml/min per 1.73 m^2 per year | -2.65 [-3.29 to -2.02] | -3.24 [-4.21 to -2.28]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Annualized eGFR slope over time was estimated by a random slopes and intercepts model using all available eGFR values adjusted on baseline Hb, region, CV history at Baseline and the interaction terms; Test type: Superiority; p = 0.316, Mixed Models Analysis; Least squares mean difference = 0.59, 95% CI 2-sided [-0.57 to 1.75]

11. Secondary Outcome: Average Level of Hb Over Weeks 28 to 36 Without Use of Rescue Therapy Within 6 Weeks Prior to and During the Evaluation Period
Description: All scheduled and unscheduled hemoglobin values from weeks 28 to 36 were taken into account for calculating the average values.
Time Frame: Weeks 28 to 36
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 311 | 139
g/dL | 11.106 [10.97 to 11.24] | 9.468 [9.29 to 9.65]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Average Level of Hb Over Weeks 28 to 36. A Mixed Model of Repeated Measures was applied using the visits over weeks 28 to 36. The results were based on the estimated difference between the two treatment arms by visit based on this MMRM model. The model included treatment arm, region, CV History, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.638, 95% CI 2-sided [1.44 to 1.84]

12. Secondary Outcome: Average Level of Hb Over Weeks 44 to 52 Without Use of Rescue Therapy Within 6 Weeks Prior to and During the Evaluation Period
Description: All scheduled and unscheduled hemoglobin values from weeks 44 to 52 were taken into account for calculating the average values.
Time Frame: Weeks 44 to 52
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 287 | 118
g/dL | 10.984 [10.85 to 11.12] | 9.381 [9.19 to 9.58]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Average Level of Hb Over Weeks 44 to 52. A Mixed Model of Repeated Measures was applied using the visits over weeks 44 to 52. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM difference p-value is for test of differences; Least squares mean difference = 1.604, 95% CI 2-sided [1.39 to 1.82]

13. Secondary Outcome: Average Level of Hb Over Weeks 96 to 104 Without Use of Rescue Therapy Within 6 Weeks Prior to and During the Evaluation Period
Description: All scheduled and unscheduled hemoglobin values from weeks 96 to 104 were taken into account for calculating the average values.
Time Frame: Weeks 96 to 104
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 120 | 32
g/dL | 10.816 [10.63 to 11.00] | 9.324 [9.01 to 9.64]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Average Level of Hb Over Weeks 96 to 104. A Mixed Model of Repeated Measures was applied using the visits over weeks 96 to 104. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.492, 95% CI 2-sided [1.14 to 1.85]

14. Secondary Outcome: Time to Achieve the First Hb Response Without Rescue Therapy, as Defined by Primary Endpoint
Description: Hb response was measured as Yes or No; Yes was defined as Hb ≥11.0 g/dL and Hb increase from baseline by ≥ 1.0 g/dL, for participants with baseline Hb > 8.0 g/dL; or Hb increase from baseline by ≥ 2.0 g/dL, for participants with baseline Hb ≤ 8.0 g/dL. For a participant without rescue therapy before Hb response (defined in 1 primary outcome), the time to achieve Hb response was calculated (in weeks) as: (First event date - Analysis date of first dose intake + 1) / 7 where First event date was defined as First date of both values that met the criteria for response. Participants who discontinued or received rescue therapy prior to the first Hb response or before the second consecutive Hb value defined as a response were classified as non responders and were censored at week 24 or end of efficacy emergent period, whichever came first. Data analysis was completed using Kaplan-Meier estimate for cumulative proportion.
Time Frame: Baseline to week 24
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
Percentage of participants
  Week 4 | 26.0 [21.6 to 30.4] | 3.5 [0.9 to 6.0]
  Week 8 | 59.8 [54.7 to 64.9] | 6.2 [2.8 to 9.7]
  Week 16 | 83.4 [79.3 to 87.5] | 9.4 [5.1 to 13.7]
  Week 24 | 89.1 [85.5 to 92.6] | 11.6 [6.8 to 16.5]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Time to Achieve the First Hb Response. Hazard ratio was calculated using stratified Cox Proportional Hazards Regression stratifying on CV history and region and adjusting on Hb and eGFR at baseline as continuous covariates; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 19.001, 95% CI 2-sided [11.98 to 30.15]

15. Secondary Outcome: Hb Change From BL to Each Post-Dosing Time Point
Description: All scheduled and unscheduled hemoglobin values that belong to each visit window were taken into account using one value per analysis window. Baseline Hb was defined as the mean of four latest central laboratory Hb values prior or on the same date as first study drug intake (pre-dose).
Time Frame: Baseline (day 1) and weeks 1, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, 100, 104
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
g/dL
  Hb Change From BL to Week 1: number analyzed (Participants) | 372 | 193
  Hb Change From BL to Week 1 | 0.390 [0.29 to 0.49] | -0.006 [-0.12 to 0.11]
  Hb Change From BL to Week 2: number analyzed (Participants) | 363 | 195
  Hb Change From BL to Week 2 | 0.977 [0.87 to 1.08] | 0.039 [-0.09 to 0.17]
  Hb Change From BL to Week 4: number analyzed (Participants) | 360 | 189
  Hb Change From BL to Week 4 | 1.591 [1.47 to 1.71] | 0.119 [-0.04 to 0.27]
  Hb Change From BL to Week 6: number analyzed (Participants) | 347 | 186
  Hb Change From BL to Week 6 | 1.927 [1.79 to 2.06] | 0.100 [-0.07 to 0.27]
  Hb Change From BL to Week 8: number analyzed (Participants) | 346 | 188
  Hb Change From BL to Week 8 | 2.236 [2.10 to 2.37] | 0.178 [0.01 to 0.35]
  Hb Change From BL to Week 10: number analyzed (Participants) | 335 | 184
  Hb Change From BL to Week 10 | 2.129 [1.99 to 2.26] | 0.180 [0.01 to 0.35]
  Hb Change From BL to Week 12: number analyzed (Participants) | 337 | 179
  Hb Change From BL to Week 12 | 2.412 [2.28 to 2.55] | 0.322 [0.15 to 0.49]
  Hb Change From BL to Week 14: number analyzed (Participants) | 332 | 174
  Hb Change From BL to Week 14 | 2.214 [2.08 to 2.35] | 0.163 [0.00 to 0.33]
  Hb Change From BL to Week 16: number analyzed (Participants) | 321 | 173
  Hb Change From BL to Week 16 | 2.365 [2.23 to 2.50] | 0.378 [0.20 to 0.56]
  Hb Change From BL to Week 18: number analyzed (Participants) | 317 | 161
  Hb Change From BL to Week 18 | 2.087 [1.95 to 2.23] | 0.246 [0.06 to 0.43]
  Hb Change From BL to Week 20: number analyzed (Participants) | 310 | 151
  Hb Change From BL to Week 20 | 2.191 [2.04 to 2.34] | 0.367 [0.18 to 0.56]
  Hb Change From BL to Week 22: number analyzed (Participants) | 312 | 149
  Hb Change From BL to Week 22 | 1.873 [1.73 to 2.02] | 0.222 [0.03 to 0.41]
  Hb Change From BL to Week 24: number analyzed (Participants) | 307 | 142
  Hb Change From BL to Week 24 | 1.802 [1.66 to 1.95] | 0.355 [0.16 to 0.55]
  Hb Change From BL to Week 28: number analyzed (Participants) | 301 | 145
  Hb Change From BL to Week 28 | 1.996 [1.85 to 2.14] | 0.435 [0.24 to 0.63]
  Hb Change From BL to Week 32: number analyzed (Participants) | 300 | 137
  Hb Change From BL to Week 32 | 1.911 [1.77 to 2.05] | 0.324 [0.13 to 0.52]
  Hb Change From BL to Week 36: number analyzed (Participants) | 290 | 131
  Hb Change From BL to Week 36 | 2.100 [1.95 to 2.25] | 0.410 [0.21 to 0.61]
  Hb Change From BL to Week 40: number analyzed (Participants) | 290 | 125
  Hb Change From BL to Week 40 | 1.887 [1.74 to 2.03] | 0.241 [0.04 to 0.45]
  Hb Change From BL to Week 44: number analyzed (Participants) | 275 | 122
  Hb Change From BL to Week 44 | 1.977 [1.82 to 2.13] | 0.278 [0.06 to 0.49]
  Hb Change From BL to Week 48: number analyzed (Participants) | 282 | 114
  Hb Change From BL to Week 48 | 1.695 [1.54 to 1.85] | 0.249 [0.03 to 0.46]
  Hb Change From BL to Week 52: number analyzed (Participants) | 267 | 111
  Hb Change From BL to Week 52 | 1.939 [1.78 to 2.10] | 0.298 [0.07 to 0.52]
  Hb Change From BL to Week 56: number analyzed (Participants) | 217 | 74
  Hb Change From BL to Week 56 | 1.725 [1.56 to 1.88] | 0.085 [-0.16 to 0.33]
  Hb Change From BL to Week 60: number analyzed (Participants) | 198 | 68
  Hb Change From BL to Week 60 | 1.988 [1.81 to 2.16] | 0.354 [0.09 to 0.62]
  Hb Change From BL to Week 64: number analyzed (Participants) | 174 | 55
  Hb Change From BL to Week 64 | 1.637 [1.45 to 1.82] | 0.233 [-0.06 to 0.52]
  Hb Change From BL to Week 68: number analyzed (Participants) | 173 | 49
  Hb Change From BL to Week 68 | 1.913 [1.74 to 2.09] | 0.414 [0.13 to 0.70]
  Hb Change From BL to Week 72: number analyzed (Participants) | 158 | 50
  Hb Change From BL to Week 72 | 1.765 [1.58 to 1.95] | 0.328 [0.03 to 0.63]
  Hb Change From BL to Week 76: number analyzed (Participants) | 156 | 47
  Hb Change From BL to Week 76 | 1.859 [1.67 to 2.05] | 0.674 [0.36 to 0.99]
  Hb Change From BL to Week 80: number analyzed (Participants) | 145 | 43
  Hb Change From BL to Week 80 | 1.752 [1.57 to 1.93] | 0.308 [0.01 to 0.61]
  Hb Change From BL to Week 84: number analyzed (Participants) | 143 | 37
  Hb Change From BL to Week 84 | 1.854 [1.66 to 2.05] | 0.480 [0.14 to 0.82]
  Hb Change From BL to Week 88: number analyzed (Participants) | 132 | 31
  Hb Change From BL to Week 88 | 1.570 [1.38 to 1.76] | 0.399 [0.06 to 0.74]
  Hb Change From BL to Week 92: number analyzed (Participants) | 125 | 32
  Hb Change From BL to Week 92 | 1.800 [1.60 to 2.00] | 0.418 [0.06 to 0.78]
  Hb Change From BL to Week 96: number analyzed (Participants) | 122 | 32
  Hb Change From BL to Week 96 | 1.701 [1.49 to 1.91] | 0.139 [-0.23 to 0.51]
  Hb Change From BL to Week 100: number analyzed (Participants) | 119 | 30
  Hb Change From BL to Week 100 | 1.763 [1.57 to 1.96] | 0.315 [-0.03 to 0.66]
  Hb Change From BL to Week 104: number analyzed (Participants) | 102 | 26
  Hb Change From BL to Week 104 | 1.857 [1.64 to 2.08] | 0.511 [0.11 to 0.91]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Hb change from BL to week 1. A Mixed Model of Repeated Measures was applied using the visits up to week 104. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 0.396, 95% CI 2-sided [0.29 to 0.50]
Statistical Analysis 2: Comparison: Roxadustat vs Placebo; Hb change from BL to week 2. A Mixed Model of Repeated Measures was applied using the visits up to Week 104. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 0.938, 95% CI 2-sided [0.81 to 1.07]
Statistical Analysis 3: Comparison: Roxadustat vs Placebo; Hb change from BL to week 4. A Mixed Model of Repeated Measures was applied using the visits up to Week 104. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.471, 95% CI 2-sided [1.30 to 1.64]
Statistical Analysis 4: Comparison: Roxadustat vs Placebo; Hb change from BL to week 6. A Mixed Model of Repeated Measures was applied using the visits up to Week 104. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.827, 95% CI 2-sided [1.64 to 2.02]
Statistical Analysis 5: Comparison: Roxadustat vs Placebo; Hb change from BL to week 8. A Mixed Model of Repeated Measures was applied using the visits up to Week 104. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 2.058, 95% CI 2-sided [1.87 to 2.25]
Statistical Analysis 6: Comparison: Roxadustat vs Placebo; Hb change from BL to week 10. A Mixed Model of Repeated Measures was applied using the visits up to Week 104. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.949, 95% CI 2-sided [1.75 to 2.14]
Statistical Analysis 7: Comparison: Roxadustat vs Placebo; Hb change from BL to week 12. A Mixed Model of Repeated Measures was applied using the visits up to Week 104. The results were based on the estimated difference between the two treatment arms by visit.The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 2.090, 95% CI 2-sided [1.90 to 2.28]
Statistical Analysis 8: Comparison: Roxadustat vs Placebo; Hb change from BL to week 14. A Mixed Model of Repeated Measures was applied using the visits up to Week 104. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 2.051, 95% CI 2-sided [1.86 to 2.24]
Statistical Analysis 9: Comparison: Roxadustat vs Placebo; Hb change from BL to week 16. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.987, 95% CI 2-sided [1.79 to 2.19]
Statistical Analysis 10: Comparison: Roxadustat vs Placebo; Hb change from BL to week 18. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.841, 95% CI 2-sided [1.64 to 2.05]
Statistical Analysis 11: Comparison: Roxadustat vs Placebo; Hb change from BL to week 20. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.824, 95% CI 2-sided [1.61 to 2.04]
Statistical Analysis 12: Comparison: Roxadustat vs Placebo; Hb change from BL to week 22. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit.The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.651, 95% CI 2-sided [1.43 to 1.87]
Statistical Analysis 13: Comparison: Roxadustat vs Placebo; Hb change from BL to week 24. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.447, 95% CI 2-sided [1.23 to 1.67]
Statistical Analysis 14: Comparison: Roxadustat vs Placebo; Hb change from BL to week 28. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.561, 95% CI 2-sided [1.34 to 1.78]
Statistical Analysis 15: Comparison: Roxadustat vs Placebo; Hb change From BL to week 32. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.587, 95% CI 2-sided [1.37 to 1.81]
Statistical Analysis 16: Comparison: Roxadustat vs Placebo; Hb Change from BL to week 36. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit.The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.690, 95% CI 2-sided [1.46 to 1.92]
Statistical Analysis 17: Comparison: Roxadustat vs Placebo; Hb change from BL to week 40. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.645, 95% CI 2-sided [1.41 to 1.88]
Statistical Analysis 18: Comparison: Roxadustat vs Placebo; Hb change from BL to week 44. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.699, 95% CI 2-sided [1.45 to 1.94]
Statistical Analysis 19: Comparison: Roxadustat vs Placebo; Hb change From BL to week 48. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.446, 95% CI 2-sided [1.20 to 1.69]
Statistical Analysis 20: Comparison: Roxadustat vs Placebo; Hb change from BL to week 52. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit.The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.641, 95% CI 2-sided [1.39 to 1.89]
Statistical Analysis 21: Comparison: Roxadustat vs Placebo; Hb change from BL to week 56. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit.The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.640, 95% CI 2-sided [1.37 to 1.91]
Statistical Analysis 22: Comparison: Roxadustat vs Placebo; Hb change from BL to week 60. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.634, 95% CI 2-sided [1.33 to 1.94]
Statistical Analysis 23: Comparison: Roxadustat vs Placebo; Hb change from BL to week 64. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.404, 95% CI 2-sided [1.08 to 1.73]
Statistical Analysis 24: Comparison: Roxadustat vs Placebo; Hb change From BL to week 68. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.499, 95% CI 2-sided [1.18 to 1.82]
Statistical Analysis 25: Comparison: Roxadustat vs Placebo; Hb change from BL to week 72. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.438, 95% CI 2-sided [1.10 to 1.78]
Statistical Analysis 26: Comparison: Roxadustat vs Placebo; Hb change from BL to week 76. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.185, 95% CI 2-sided [0.83 to 1.54]
Statistical Analysis 27: Comparison: Roxadustat vs Placebo; Hb change from BL to week 80. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.443, 95% CI 2-sided [1.11 to 1.78]
Statistical Analysis 28: Comparison: Roxadustat vs Placebo; Hb change from BL to week 84. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.374, 95% CI 2-sided [0.99 to 1.75]
Statistical Analysis 29: Comparison: Roxadustat vs Placebo; Hb change from BL to week 88. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.171, 95% CI 2-sided [0.79 to 1.55]
Statistical Analysis 30: Comparison: Roxadustat vs Placebo; Hb change from BL to week 92. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.382, 95% CI 2-sided [0.98 to 1.78]
Statistical Analysis 31: Comparison: Roxadustat vs Placebo; Hb change from BL to week 96. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.563, 95% CI 2-sided [1.15 to 1.97]
Statistical Analysis 32: Comparison: Roxadustat vs Placebo; Hb change from BL to week 100. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.448, 95% CI 2-sided [1.06 to 1.83]
Statistical Analysis 33: Comparison: Roxadustat vs Placebo; Hb change from BL to week 104. A Mixed Model of Repeated Measures was applied. The results were based on the estimated difference between the two treatment arms by visit. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.347, 95% CI 2-sided [0.90 to 1.79]

16. Secondary Outcome: Hb Change From BL to the Average Hb Value of Weeks 28-36 Regardless of the Use of Rescue Therapy
Description: The Hb values from visit windows from weeks 28 to 36 were used for the calculation of the average regardless of rescue therapy. Baseline Hb was defined as the mean of four latest central laboratory Hb values prior or on the same date as first study drug intake (pre-dosing).
Time Frame: Baseline and weeks 28 to 36
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 312 | 146
g/dL | 2.013 [1.88 to 2.15] | 0.399 [0.22 to 0.58]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Change from baseline to average Hb weeks 28-36. A Mixed Model of Repeated Measures was applied using the visits up to week 36. The results were based on the estimated difference between the two treatment arms overall mean effect during week 28 to 36 period based on this MMRM model. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM difference p-value is for test of differences; Least squares mean difference = 1.614, 95% CI 2-sided [1.42 to 1.81]

17. Secondary Outcome: Hb Change From BL to the Average Hb Value of Weeks 44-52 Regardless of the Use of Rescue Therapy
Description: The Hb values from visit windows from weeks 44 to 52 were used for the calculation of the average regardless of rescue therapy. Baseline Hb was defined as the mean of four latest central laboratory Hb values prior or on the same date as first study drug intake (pre-dosing).
Time Frame: Baseline and weeks 44 to 52
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 291 | 123
g/dL | 1.886 [1.75 to 2.03] | 0.292 [0.10 to 0.48]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Change from baseline to average Hb weeks 44-52. A Mixed Model of Repeated Measures was applied using the visits up to week 52. The results were based on the estimated difference between the two treatment arms overall mean effect during week 44 to 52 period based on this MMRM model. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 1.594, 95% CI 2-sided [1.38 to 1.81]

18. Secondary Outcome: Hb Change From BL to the Average Hb Value of Weeks 96-104 Regardless of the Use of Rescue Therapy
Description: The Hb values from visit windows from weeks 96 to 104 were used for the calculation of the average regardless of rescue therapy. Baseline Hb was defined as the mean of four latest central laboratory Hb values prior or on the same date as first study drug intake (pre-dosing).
Time Frame: Baseline and weeks 96 to 104
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 124 | 32
g/dL | 1.779 [1.60 to 1.96] | 0.327 [0.01 to 0.64]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Change from BL to average Hb weeks 96-104. A Mixed Model of Repeated Measures was applied using the visits up to week 104. The results were based on the estimated difference between the two treatment arms overall mean effect during week 96 to 104 period based on this MMRM model. The model included treatment arm, region, CV history, visits and visit by treatment as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — LSM difference p-value is for test of differences; Least squares mean difference = 1.452, 95% CI 2-sided [1.10 to 1.80]

19. Secondary Outcome: Percentage of Hb Values Within 10.0-12.0 g/dL in Weeks 28-36 Without Use of Rescue Therapy
Description: The percentage of Hb values measured during weeks 28-36 within 10.0 -12.0 g/dL, without having received rescue therapy within 6 weeks prior to and during the 8-week evaluation period is reported.
Time Frame: Baseline and weeks 28 to 36
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of Hb values
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 311 | 139
Percentage of Hb values | 64.18 (32.90) | 34.20 (39.47)

20. Secondary Outcome: Percentage of Hb Values Within 10.0-12.0 g/dL in Weeks 44-52 Without Use of Rescue Therapy
Description: The percentage of Hb values measured during weeks 44-52 with values within 10.0 - 12.0 g/dL, without having received rescue therapy within 6 weeks prior to and during the 8-week evaluation period is reported.
Time Frame: Baseline and weeks 44 to 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of Hb values
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 287 | 118
Percentage of Hb values | 69.39 (32.47) | 35.45 (41.75)

21. Secondary Outcome: Percentage of Hb Values Within 10.0-12.0 g/dL in Weeks 96-104 Without Use of Rescue Therapy
Description: The percentage of Hb values measured during weeks 96-104 within 10.0 -12.0 g/dL, without having received rescue therapy within 6 weeks prior to and during the 8-week evaluation period is reported.
Time Frame: Baseline and weeks 96 to 104
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of Hb values
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 120 | 32
Percentage of Hb values | 64.65 (37.16) | 40.63 (44.39)

22. Secondary Outcome: Time to First Hospitalization
Description: Time to first hospitalization was defined in years as the First event date during the Efficacy Emergent Period - (Analysis date of first dose intake +1)/365.25. The first event date was defined as the Date of first admission. The Efficacy Emergent Period was defined as the evaluation period from the analysis date of first dose intake up to 7 days after the analysis date of last dose or EOT visit, whichever occured first. Analysis date of first dose intake was defined as the date of first study drug intake collected on day 1 visit. For participants who experienced more than one hospitalization, only their first event following study treatment was used. Data analysis was completed using Kaplan-Meier estimate for cumulative proportion.
Time Frame: Baseline to week 104
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
Percentage of participants
  Year 0.5 | 32.2 [27.3 to 37.0] | 39.8 [32.7 to 46.9]
  Year 1 | 49.9 [44.6 to 55.2] | 49.3 [41.8 to 56.8]
  Year 1.5 | 62.1 [56.3 to 67.9] | 64.0 [54.5 to 73.4]
  Year 2 | NA [NA to NA] — Due to low number of events estimate for this time point could not be calculated. | 67.8 [57.9 to 77.7]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.643, Regression, Cox; Hazard Ratio (HR) = 0.945, 95% CI 2-sided [0.74 to 1.20]

23. Secondary Outcome: Number of Days of Hospitalization Per Patient Exposure Year (PEY)
Description: The sum of the durations of all hospitalizations in days was adjusted for the duration of exposure. Derived only for participants with at least one hospitalization. The number of days of hospitalization per PEY was calculated as the sum of the durations of all hospitalizations in days [Minimum (Date of discharge, End of Efficacy Emergent Period) - Date of admission + 1] / [Duration of Efficacy Emergent Period in days / 365.25]. Participants can have more than one hospitalization.
Time Frame: Baseline to week 104
Population: The analysis population was the FAS, which consisted of participants with hospitalizations.
Measure: Mean (Standard Deviation); unit: Number of days per PEY
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
Number of days per PEY | 14.567 (29.214) | 15.885 (30.224)

24. Secondary Outcome: Time to First Use of Rescue Therapy (Composite of RBC, Transfusions, ESA Use, and IV Iron) in the First 24 Weeks of Treatment
Description: Time to first use of rescue therapy in years. Data analysis was completed using Kaplan-Meier estimate for cumulative proportion.
Time Frame: Baseline to week 24
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
Percentage of participants
  Week 6 | 0.8 [0.0 to 1.7] | 6.0 [2.7 to 9.3]
  Week 12 | 2.5 [0.9 to 4.1] | 15.8 [10.7 to 20.9]
  Week 18 | 3.3 [1.5 to 5.2] | 25.3 [19.2 to 31.5]
  Week 24 | 5.5 [3.1 to 7.9] | 32.1 [25.4 to 38.7]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Time to start rescue therapy within first 24 weeks. Hazard ratio was calculated using stratified Cox Proportional Hazards Regression stratifying on CV history and region and adjusting on Hb and eGFR at baseline as continuous covariates; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.139, 95% CI 2-sided [0.08 to 0.23]

25. Secondary Outcome: Time to First Use of RBC Transfusions
Description: Time to First Use of RBC Transfusions during efficacy emergent period. For participants who have experienced more than one RBC transfusion, only their first event following study treatment was used. The efficacy emergent period was defined as the evaluation period from the analysis date of first dose intake up to 7 days after the analysis date of last dose or EOT visit, whichever occured first. Data analysis was completed using Kaplan-Meier estimate for cumulative proportion.
Time Frame: Baseline to week 104
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
Percentage of participants
  Year 0.5 | 2.9 [1.1 to 4.7] | 15.2 [10.1 to 20.4]
  Year 1 | 5.6 [3.0 to 8.1] | 20.2 [14.2 to 26.2]
  Year 1.5 | 12.1 [7.7 to 16.5] | 21.8 [15.1 to 28.5]
  Year 2 | 15.0 [9.9 to 20.1] | 27.0 [17.7 to 36.4]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p < 0.001, Regression, Cox; Cox Proportional Hazard = 0.343, 95% CI 2-sided [0.21 to 0.55]

26. Secondary Outcome: Mean Monthly Number of RBC Packs
Description: During efficacy emergent period, the mean monthly number of RBC packs was calculated as the sum of units transfused between the first dose and up to the last dose in the period divided by duration of efficacy emergent period (in days) divided by 28 days. The efficacy emergent period was defined as the evaluation period from the analysis date of first dose intake up to 7 days after the analysis date of last dose or EOT visit, whichever occured first. In case of missing number of packs, values were estimated based on 1 unit for packed cells = 250 mL or 1 unit for whole blood = 500 mL. Participants without RBC transfusion were included with a value of zero. No estimation if values were missing.
Time Frame: Baseline to week 104
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: RBC Packs per 28 days
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
RBC Packs per 28 days | 0.041 (0.397) | 0.089 (0.243)
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; The Analysis of Covariance (ANCOVA) model was applied including treatment as fixed factor, region and history of CV disease as class factors and baseline Hb, baseline eGFR as continuous covariates; Test type: Superiority; p = 0.128, ANCOVA; Least squares mean difference = -0.045, 95% CI 2-sided [-0.10 to 0.01]

27. Secondary Outcome: Mean Monthly Volume of Blood Transfused
Description: During efficacy emergent period, the mean monthly volume of blood transfused was calculated as the sum of blood volume transfused between the first dose and up to the last dose in the period divided by duration of efficacy emergent period (in days) divided by 28 days. The efficacy emergent period was defined as the evaluation period from the analysis date of first dose intake up to 7 days after the analysis date of last dose or EOT visit, whichever occurred first. The mean monthly volume transfused was calculated as the sum of the volume transfused between the first dose and up to the last dose in the period divided by duration (in days) and multiplied by 28 days. Participants without RBC transfusion were included with a value of zero.
Time Frame: Baseline to week 104
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Milliliters (ml) per 28 days
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
Milliliters (ml) per 28 days | 11.331 (106.624) | 22.596 (60.666)
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; The Analysis of Covariance (ANCOVA) model was applied included treatment arm, region, CV history as categorical variables and baseline Hb and baseline eGFR as continuous variables; Test type: Superiority; p = 0.183, ANCOVA; Least squares mean difference = -10.429, 95% CI 2-sided [-25.81 to 4.95]

28. Secondary Outcome: Time to First Use of ESA Rescue Therapy
Description: Time to First Use of ESA Rescue Therapy during efficacy emergent period. For participants with use of ESA, the time to first use of ESA was calculated as (First event date - Analysis date of first dose intake + 1) / 365.25. The efficacy emergent period was defined as the evaluation period from the analysis date of first dose intake up to 7 days after the analysis date of last dose or EOT visit, whichever occured first. Data analysis was completed using Kaplan-Meier estimate for cumulative proportion. Participants without ESA rescue were censored at the end of treatment.
Time Frame: Baseline to week 104
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
Percentage of participants
  Year 0.5 | 1.8 [0.4 to 3.2] | 20.4 [14.5 to 26.3]
  Year 1 | 4.8 [2.4 to 7.2] | 36.4 [28.9 to 43.9]
  Year 1.5 | 6.0 [3.1 to 8.9] | 42.3 [33.9 to 50.8]
  Year 2 | 6.7 [3.5 to 9.9] | 42.3 [33.9 to 50.8]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.101, 95% CI 2-sided [0.06 to 0.17]

29. Secondary Outcome: Time to First Use of IV Iron
Description: Time to first use of IV iron during efficacy emergent period in years. For participants with use of IV iron, the time to first use of IV iron was calculated as (First event date - Analysis date of first dose intake + 1) / 365.25. The efficacy emergent period was defined as the evaluation period from the analysis date of first dose intake up to 7 days after the analysis date of last dose or EOT visit, whichever occurred first.Data analysis was completed using Kaplan-Meier estimate for cumulative proportion.
Time Frame: Baseline to week 104
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
Percentage of participants
  Year 0.5 | 2.3 [0.7 to 3.9] | 6.2 [2.7 to 9.8]
  Year 1 | 5.3 [2.8 to 7.8] | 9.4 [4.8 to 14.0]
  Year 1.5 | 7.5 [4.3 to 10.7] | 10.7 [5.5 to 15.9]
  Year 2 | 10.6 [6.3 to 14.8] | 19.1 [8.8 to 29.5]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.045, Regression, Cox; Hazard Ratio (HR) = 0.538, 95% CI 2-sided [0.29 to 0.99]

30. Secondary Outcome: Change From BL to Each Post-Dosing Visit in Total Cholesterol
Description: Change from baseline to each planned assessment for total cholesterol is reported. Baseline was defined as the value on day 1. If the value was missing, the latest value prior to first study drug administration was used.
Time Frame: Baseline and weeks 4, 8, 12, 20, 28, 36, 44, 52, 68, 84, 104
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
mmol/L
  Week 4: number analyzed (Participants) | 368 | 194
  Week 4 | -1.151 (1.058) | 0.108 (0.842)
  Week 8: number analyzed (Participants) | 348 | 191
  Week 8 | -1.066 (1.086) | 0.048 (0.932)
  Week 12: number analyzed (Participants) | 342 | 185
  Week 12 | -0.836 (1.173) | 0.088 (1.116)
  Week 20: number analyzed (Participants) | 323 | 167
  Week 20 | -0.747 (1.227) | 0.193 (1.129)
  Week 28: number analyzed (Participants) | 310 | 149
  Week 28 | -0.816 (1.284) | 0.201 (1.271)
  Week 36: number analyzed (Participants) | 295 | 133
  Week 36 | -0.803 (1.300) | 0.183 (1.174)
  Week 44: number analyzed (Participants) | 285 | 126
  Week 44 | -0.854 (1.238) | 0.077 (1.346)
  Week 52: number analyzed (Participants) | 278 | 120
  Week 52 | -0.815 (1.314) | 0.104 (1.304)
  Week 68: number analyzed (Participants) | 197 | 67
  Week 68 | -0.971 (1.382) | 0.188 (1.222)
  Week 84: number analyzed (Participants) | 154 | 43
  Week 84 | -1.055 (1.554) | 0.102 (1.284)
  Week 104: number analyzed (Participants) | 123 | 32
  Week 104 | -0.944 (1.584) | 0.218 (1.067)

31. Secondary Outcome: Change From BL to Each Post-Dosing Visit in Low Density Lipoprotein (LDL)/High-Density Lipoprotein (HDL) Ratio
Description: Change from baseline to each planned assessment for LDL/HDL ratio is reported. Baseline was defined as the value on Day 1. If this value was missing, the latest value prior to first study drug administration was used.
Time Frame: Baseline and weeks 4, 8, 12, 20, 28, 36, 44, 52, 68, 84, 104
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
Ratio
  Week 4: number analyzed (Participants) | 367 | 193
  Week 4 | -0.331 (0.777) | 0.076 (0.635)
  Week 8: number analyzed (Participants) | 347 | 190
  Week 8 | -0.374 (0.952) | 0.068 (0.685)
  Week 12: number analyzed (Participants) | 341 | 185
  Week 12 | -0.268 (0.905) | 0.081 (0.915)
  Week 20: number analyzed (Participants) | 322 | 166
  Week 20 | -0.250 (1.024) | 0.155 (0.788)
  Week 28: number analyzed (Participants) | 309 | 149
  Week 28 | -0.313 (1.057) | 0.156 (0.861)
  Week 36: number analyzed (Participants) | 293 | 133
  Week 36 | -0.349 (1.040) | 0.157 (1.053)
  Week 44: number analyzed (Participants) | 283 | 126
  Week 44 | -0.368 (1.099) | 0.099 (1.198)
  Week 52: number analyzed (Participants) | 277 | 120
  Week 52 | -0.429 (1.125) | 0.019 (1.076)
  Week 68: number analyzed (Participants) | 196 | 67
  Week 68 | -0.466 (1.219) | 0.052 (0.955)
  Week 84: number analyzed (Participants) | 154 | 43
  Week 84 | -0.509 (1.307) | 0.114 (1.113)
  Week 104: number analyzed (Participants) | 122 | 32
  Week 104 | -0.414 (1.306) | 0.105 (0.873)

32. Secondary Outcome: Change From BL to Each Post-Dosing Visit in Non-HDL Cholesterol
Description: Change from baseline to each planned assessment for non-HDL is reported. Baseline was defined as the value on day 1. If this value was missing, the latest value prior to first study drug administration was used.
Time Frame: Baseline and weeks 4, 8, 12, 20, 28, 36, 44, 52, 68, 84, 104
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
mmol/L
  Week 4: number analyzed (Participants) | 367 | 193
  Week 4 | -0.969 (0.989) | 0.118 (0.789)
  Week 8: number analyzed (Participants) | 347 | 190
  Week 8 | -0.909 (1.064) | 0.070 (0.864)
  Week 12: number analyzed (Participants) | 341 | 185
  Week 12 | -0.709 (1.107) | 0.078 (1.050)
  Week 20: number analyzed (Participants) | 322 | 166
  Week 20 | -0.638 (1.175) | 0.186 (1.072)
  Week 28: number analyzed (Participants) | 309 | 149
  Week 28 | -0.710 (1.227) | 0.206 (1.227)
  Week 36: number analyzed (Participants) | 293 | 133
  Week 36 | -0.711 (1.239) | 0.202 (1.133)
  Week 44: number analyzed (Participants) | 283 | 125
  Week 44 | -0.751 (1.190) | 0.106 (1.342)
  Week 52: number analyzed (Participants) | 277 | 120
  Week 52 | -0.751 (1.276) | 0.104 (1.299)
  Week 68: number analyzed (Participants) | 196 | 67
  Week 68 | -0.882 (1.325) | 0.174 (1.187)
  Week 84: number analyzed (Participants) | 154 | 43
  Week 84 | -0.939 (1.518) | 0.089 (1.343)
  Week 104: number analyzed (Participants) | 123 | 32
  Week 104 | -0.839 (1.554) | 0.174 (1.014)

33. Secondary Outcome: Change From BL to Each Post-Dosing Visit in Apolipoproteins A1 (ApoA1)
Description: Change from baseline to each planned assessment for apolipoproteins A1 is reported. Baseline was defined as the value on day 1. If this value was missing, the latest value prior to first study drug administration was used.
Time Frame: Baseline and weeks 4, 8, 12, 20, 28, 36, 44, 52, 68, 84, 104
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 188 | 105
g/L
  Week 4: number analyzed (Participants) | 183 | 102
  Week 4 | -0.168 (0.232) | 0.013 (0.190)
  Week 8: number analyzed (Participants) | 174 | 102
  Week 8 | -0.148 (0.229) | 0.008 (0.227)
  Week 12: number analyzed (Participants) | 170 | 97
  Week 12 | -0.131 (0.254) | 0.004 (0.203)
  Week 20: number analyzed (Participants) | 158 | 90
  Week 20 | -0.114 (0.245) | 0.036 (0.222)
  Week 28: number analyzed (Participants) | 134 | 67
  Week 28 | -0.104 (0.265) | 0.006 (0.233)
  Week 36: number analyzed (Participants) | 149 | 77
  Week 36 | -0.101 (0.252) | 0.002 (0.223)
  Week 44: number analyzed (Participants) | 140 | 72
  Week 44 | -0.135 (0.259) | -0.013 (0.268)
  Week 52: number analyzed (Participants) | 139 | 71
  Week 52 | -0.090 (0.260) | -0.028 (0.248)
  Week 68: number analyzed (Participants) | 63 | 28
  Week 68 | -0.157 (0.310) | 0.018 (0.204)
  Week 84: number analyzed (Participants) | 30 | 12
  Week 84 | -0.132 (0.282) | 0.060 (0.196)
  Week 104: number analyzed (Participants) | 12 | 4
  Week 104 | -0.098 (0.227) | 0.070 (0.136)

34. Secondary Outcome: Change From BL to Each Post-Dosing Visit in Apolipoproteins B (ApoB)
Description: Change from baseline to each planned assessment for apolipoproteins B is reported. Baseline was defined as the value on day 1. If this value was missing, the latest value prior to first study drug administration was used.
Time Frame: Baseline and weeks 4, 8, 12, 20, 28, 36, 44, 52, 68, 84, 104
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 188 | 105
mg/dL
  Week 4: number analyzed (Participants) | 183 | 102
  Week 4 | -19.891 (20.669) | 2.059 (22.220)
  Week 8: number analyzed (Participants) | 174 | 102
  Week 8 | -19.483 (21.009) | 2.059 (20.297)
  Week 12: number analyzed (Participants) | 170 | 97
  Week 12 | -14.935 (24.613) | 0.278 (21.707)
  Week 20: number analyzed (Participants) | 158 | 90
  Week 20 | -12.709 (24.424) | 5.711 (25.883)
  Week 28: number analyzed (Participants) | 133 | 67
  Week 28 | -13.782 (28.634) | 9.746 (26.864)
  Week 36: number analyzed (Participants) | 149 | 77
  Week 36 | -14.866 (25.469) | 6.623 (25.895)
  Week 44: number analyzed (Participants) | 140 | 72
  Week 44 | -15.593 (26.594) | 3.222 (30.771)
  Week 52: number analyzed (Participants) | 139 | 71
  Week 52 | -14.122 (27.503) | 4.676 (31.440)
  Week 68: number analyzed (Participants) | 63 | 28
  Week 68 | -18.746 (28.633) | 2.786 (28.900)
  Week 84: number analyzed (Participants) | 30 | 12
  Week 84 | -20.133 (28.134) | 12.500 (32.152)
  Week 104: number analyzed (Participants) | 12 | 4
  Week 104 | -10.917 (22.885) | 14.750 (20.271)

35. Secondary Outcome: Change From BL to Each Post-Dosing Visit in Ratio ApoB/ApoA1
Description: Change from baseline to each planned assessment for ratio of ApoB/ApoA1 is reported. Baseline was defined as the value on day 1. If this value was missing, the latest value prior to first study drug administration was used.
Time Frame: Baseline and weeks 4, 8, 12, 20, 28, 36, 44, 52, 68, 84, 104
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
Ratio
  Week 4: number analyzed (Participants) | 183 | 101
  Week 4 | -0.073 (0.165) | 0.010 (0.169)
  Week 8: number analyzed (Participants) | 172 | 101
  Week 8 | -0.084 (0.202) | 0.000 (0.184)
  Week 12: number analyzed (Participants) | 169 | 96
  Week 12 | -0.059 (0.164) | -0.006 (0.201)
  Week 20: number analyzed (Participants) | 158 | 89
  Week 20 | -0.043 (0.189) | 0.009 (0.198)
  Week 28: number analyzed (Participants) | 133 | 66
  Week 28 | -0.066 (0.222) | 0.063 (0.205)
  Week 36: number analyzed (Participants) | 149 | 76
  Week 36 | -0.070 (0.200) | 0.045 (0.213)
  Week 44: number analyzed (Participants) | 140 | 71
  Week 44 | -0.053 (0.220) | 0.031 (0.265)
  Week 52: number analyzed (Participants) | 137 | 70
  Week 52 | -0.065 (0.207) | 0.047 (0.266)
  Week 68: number analyzed (Participants) | 63 | 28
  Week 68 | -0.086 (0.212) | 0.001 (0.184)
  Week 84: number analyzed (Participants) | 29 | 12
  Week 84 | -0.066 (0.210) | 0.058 (0.295)
  Week 104: number analyzed (Participants) | 12 | 4
  Week 104 | -0.024 (0.126) | 0.085 (0.132)

36. Secondary Outcome: Percentage of Participants With Mean LDL Cholesterol <100 mg/dL Calculated Over Weeks 12 to 28
Description: Mean LDL cholesterol <100 mg/dL over weeks 12 to 28 was defined as a binary variable (Yes/No), where Yes was defined as mean LDL cholesterol <100 mg/dL over weeks 12 to 28. Participants without any LDL value within this duration were excluded.
Time Frame: Weeks 12 to 28
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
Percentage of Participants
  Yes (Regardless of fasting status) | 62.9 | 41.1
  No (Regardless of fasting status) | 37.1 | 58.9

37. Secondary Outcome: Percentage of Participants Who Have Achieved Antihypertensive Treatment Goal in CKD Participants Over Weeks 12-28
Description: Occurrence of achieved antihypertensive treatment goal was defined as the average SBP < 130 mmHg and the average DBP < 80 mmHg over the period of weeks 12-28. Participants without any blood pressure measurement were excluded.
Time Frame: Weeks 12 to 28
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
Percentage of Participants
  Yes | 25.6 | 28.0
  No | 74.4 | 72.0

38. Secondary Outcome: Change From BL to the Average Value of Weeks 12-28 in Quality of Life (QoL) SF-36 Physical Component Score (PCS)
Description: The 36-Item short-form health survey (SF-36) is a multi-purpose survey with 36 questions. It provides an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures. For each scale scores range from 0-100. The physical component score was calculated based on the results of the SF-36 scores. Higher scores indicate better health status.
Time Frame: Baseline and weeks 12 to 28
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 340 | 185
Units on a Scale | 1.842 [0.88 to 2.80] | 1.468 [0.34 to 2.59]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; The Mixed Model of Repeated Measures included treatment, visit (week 8, week 12 and week 28), visit by treatment interaction, region and history of CV disease as fixed class factors and baseline SF-36 PCS, baseline Hb, baseline eGFR as continuous covariates; Test type: Superiority; p = 0.475, Mixed Models Analysis — LSM Difference p-value is for test of differences; Least squares mean difference = 0.374, 95% CI 2-sided [-0.65 to 1.40]

39. Secondary Outcome: Change From BL to the Average Value of Weeks 12-28 in Anemia Subscale (Ans) of Functional Assessment of Cancer Therapy (FACT-An) Score
Description: Baseline FACT-An AnS was defined as the FACT-An AnS value on Day 1. Together with the Functional Assessment of Cancer Therapy - General (FACT-G), the Anemia Subscale (AnS) is referred to as the FACT-An Total. The AnS scale contains 13 fatigue specific items (the Fatigue Score) plus 7 items related to anemia. The Anemia AnS score range is 0 to 80. For the above score, a higher score indicates better QoL.
Time Frame: Baseline and weeks 12 to 28
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 339 | 185
Units on a Scale | 4.470 [2.86 to 6.08] | 2.766 [0.91 to 4.62]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; A Mixed Model of Repeated Measures was applied using the visits up to week 28. The model includes treatment, visit (week 8, week 12 and week 28), visit by treatment interaction, region and history of CV disease as fixed class factors and baseline FACT-An Ans, baseline Hb, baseline eGFR as continuous covariates. Baseline FACT-An Ans is defined as the FACT-An Ans value on day 1; Test type: Superiority; p = 0.047, Mixed Models Analysis — LSM difference p-value is for test of differences; Least squares mean difference = 1.704, 95% CI 2-sided [0.02 to 3.38]

40. Secondary Outcome: Change From BL to the Average Value of Weeks 12-28 in Total FACT-An Score
Description: Baseline FACT-An Total Score was defined as the FACT-An Total score on Day 1. Total Fact-An score is composed of FACT-G and Ans scales. FACT-G contains 27 items that cover four dimensions of well-being: physical (PWB) - 7 items, functional (FWB) - 7 items, social/family (SWB) - 7 items, and emotional (EWB) - 6 items. The AnS scale contains 13 fatigue specific items (the Fatigue Score) plus 7 items related to anemia. The total score is obtained by summation of the scores from PWB, SWB, EWB, FWB and AnS. The FACT-An Total Score scale range is 0-188. A higher score indicates better QoL.
Time Frame: Baseline and weeks 12 to 28
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 338 | 185
Units on a Scale | 5.777 [2.60 to 8.95] | 3.691 [0.01 to 7.37]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; A Mixed Model of Repeated Measures was applied using the visits up to week 28. The results were based on the estimated difference between the two treatment arms overall mean effect during week 12 to 28 period based on this MMRM model.The model includes treatment, visit (week8, week12 and week28), visit by treatment interaction, region and history of CV disease as fixed class factors and baseline FACT-An Total Score, baseline Hb, baseline eGFR as continuous covariates; Test type: Superiority; p = 0.225, Mixed Models Analysis; Least squares mean difference = 2.086, 95% CI 2-sided [-1.29 to 5.46]

41. Secondary Outcome: Change From BL to the Average Value of Weeks 12-28 in the Euroqol Questionnaire - 5 Dimensions 5 Levels (EQ-5D 5L) Visual Analogue Scale (VAS) Score
Description: The Euroqol Questionnaire - 5 Dimensions 5 Levels (EQ-5D 5L) is a self-reported questionnaire. The EQ-5D 5L is used as a measure of respondents' Health Related Quality of Life (HRQoL). The EQ-5D 5L consists of the EQ-5D descriptive system and the EQ visual analogue scale (VAS). The EQ-5D 5L descriptive system comprises of 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, extreme problems. The VAS records the respondent's self-rated health status on a graduated (0-100) scale, where the answers are labeled 'Best imaginable health state' and 'Worst imaginable health state' with higher scores for higher HRQoL.
Time Frame: Baseline and weeks 12 to 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 340 | 184
Units on a Scale | 5.390 (17.278) | 0.990 (15.859)

42. Secondary Outcome: Change From BL to the Average Value of Weeks 12-28 in Overall Work Impairment Due to Anaemic Symptoms
Description: Work productivity and activity impairment: anemic symptoms (WPAI:ANS) questionnaire version 2 was used to measure work and activity impairment during the last seven days due to anemia. It is self-assessed questionnaire which consists of 6 questions covering work and daily activities. Questions include asking if participant is working, how many hours the person missed work due to anemic symptoms, how many hours the person missed work due to other reasons, how many hours participant actually worked and how the anemic symptoms impacted their productivity and ability to do daily activities. For the last 2 questions, they were scored from 0-10 with 0 identifying no effect on work and 10 completely prevented from working. Overall work impairment due to ANS was calculated as 100 x Q2/(Q2+Q4)+[(1-Q2/(Q2+Q4))x(Q5/10)]. Scores were calculated with the formula to derive the overall work impairment on each timepoints in percentage, and then changes of the percentage from baseline are reported.
Time Frame: Baseline and weeks 12 to 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of work impairment
Groups:
- Placebo: Participants received matching placebo according to the tiered weight-based approach, with starting doses of 70 mg given thrice weekly (TIW) to participants weighing up to 70 kg and 100 mg given TIW to participants weighing more than 70 kg. Dose-titration was performed based upon regular measurement of Hb levels until participants achieved central Hb value of ≥ 11.0 g/dL and Hb increase from baseline (BL) of ≥ 1.0 g/dL at two consecutive study visits, separated by at least 5 days. Once target Hb level was reached participants entered maintenance period during which roxadustat dosage was adjusted every 4 weeks to maintain participants Hb level within the target range of 10.0 g/dL and 12.0 g/dL. Participants received matching placebo for at least 52 weeks up to a maximum of 104 weeks.Participants were treated with placebo three times a week (TIW) for at least 52 weeks up to a maximum of 104 weeks. Treatment dosage was adjusted based on the predefined targeted hemoglobin (Hb) values.
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
Percentage of work impairment | -5.965 (21.856) | -4.230 (23.679)

43. Secondary Outcome: Percentage of Participants in Each Category in Patients' Global Impression of Change (PGIC)
Description: The Patients' Global Impression of Change (PGIC) is a participant-rated instrument that measures change in participants overall status on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: Week 12 to 28
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
Percentage of Participants
  Week 12 [Very much improved + Much improved] | 41.2 | 18.9
  Week 28 [Very much improved + Much improved] | 46.4 | 28.6

44. Secondary Outcome: Change From BL to Each Study Visit in Serum Hepcidin
Description: Baseline was assessed on Day 1 visit. If baseline value was missing, the value from screening visit was used. In case of missing data, no imputation rules were applied.
Time Frame: Baseline and weeks 4,12,20,36,52,104
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 382 | 195
ug/L
  Week 4: number analyzed (Participants) | 345 | 182
  Week 4 | -19.835 (29.765) | 1.748 (35.368)
  Week 12: number analyzed (Participants) | 323 | 171
  Week 12 | -17.369 (31.572) | 0.971 (33.952)
  Week 20: number analyzed (Participants) | 303 | 148
  Week 20 | -10.684 (35.858) | -1.879 (30.661)
  Week 36: number analyzed (Participants) | 218 | 98
  Week 36 | -12.981 (32.351) | 0.803 (39.816)
  Week 52: number analyzed (Participants) | 268 | 114
  Week 52 | -12.274 (37.445) | 2.025 (40.678)
  Week 104: number analyzed (Participants) | 108 | 28
  Week 104 | -10.051 (33.671) | -7.436 (22.923)

45. Secondary Outcome: Change From BL to Each Study Visit in Serum Ferritin
Description: Baseline assessment was assessment from Day 1 visit. If baseline value was missing, the value from screening visit was used. In case of missing data, no imputation rules were applied.
Time Frame: Baseline and weeks 4, 8, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 104
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
pmol/L
  Week 4: number analyzed (Participants) | 360 | 192
  Week 4 | -221.827 (248.902) | 11.564 (335.096)
  Week 8: number analyzed (Participants) | 346 | 191
  Week 8 | -247.955 (295.920) | 1.789 (309.673)
  Week 12: number analyzed (Participants) | 337 | 179
  Week 12 | -265.812 (318.433) | -21.098 (254.782)
  Week 20: number analyzed (Participants) | 318 | 154
  Week 20 | -198.349 (284.015) | -32.561 (320.382)
  Week 28: number analyzed (Participants) | 308 | 146
  Week 28 | -184.501 (341.114) | -5.123 (470.691)
  Week 36: number analyzed (Participants) | 295 | 132
  Week 36 | -142.876 (608.677) | 36.005 (538.357)
  Week 44: number analyzed (Participants) | 287 | 124
  Week 44 | -137.151 (352.715) | 57.373 (594.125)
  Week 52: number analyzed (Participants) | 276 | 118
  Week 52 | 164.009 (564.396) | 93.245 (640.998)
  Week 60: number analyzed (Participants) | 200 | 70
  Week 60 | -133.499 (467.931) | -18.833 (441.131)
  Week 68: number analyzed (Participants) | 177 | 50
  Week 68 | -159.906 (453.802) | 39.794 (581.616)
  Week 76: number analyzed (Participants) | 160 | 47
  Week 76 | -149.226 (408.126) | 25.291 (627.834)
  Week 84: number analyzed (Participants) | 149 | 38
  Week 84 | -103.284 (530.021) | 93.647 (753.265)
  Week 92: number analyzed (Participants) | 132 | 32
  Week 92 | -106.070 (464.192) | 1.011 (474.434)
  Week 100: number analyzed (Participants) | 127 | 30
  Week 100 | -119.647 (452.209) | 30.829 (514.823)
  Week 104: number analyzed (Participants) | 112 | 30
  Week 104 | -107.814 (458.702) | 4.524 (475.524)

46. Secondary Outcome: Change From BL to Each Study Visit in Serum Transferrin Saturation (TSAT)
Description: as for outcome 44
Time Frame: Baseline and weeks 4, 8, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 104
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage saturated
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
Percentage saturated
  Week 4: number analyzed (Participants) | 357 | 190
  Week 4 | -7.4 (11.7) | 0.7 (11.4)
  Week 8: number analyzed (Participants) | 344 | 191
  Week 8 | -5.7 (11.7) | -0.4 (13.0)
  Week 12: number analyzed (Participants) | 334 | 181
  Week 12 | -4.6 (13.5) | -0.7 (11.5)
  Week 20: number analyzed (Participants) | 317 | 152
  Week 20 | -1.1 (13.4) | -0.3 (11.5)
  Week 28: number analyzed (Participants) | 306 | 145
  Week 28 | -1.8 (13.8) | 0.8 (13.2)
  Week 36: number analyzed (Participants) | 292 | 127
  Week 36 | -1.6 (13.6) | 1.1 (14.6)
  Week 44: number analyzed (Participants) | 281 | 123
  Week 44 | -0.2 (14.0) | 1.0 (16.0)
  Week 52: number analyzed (Participants) | 275 | 115
  Week 52 | -0.7 (13.6) | 0.0 (16.3)
  Week 60: number analyzed (Participants) | 198 | 68
  Week 60 | -0.6 (14.1) | -2.7 (13.9)
  Week 68: number analyzed (Participants) | 177 | 49
  Week 68 | -2.2 (13.1) | -3.3 (12.3)
  Week 76: number analyzed (Participants) | 158 | 44
  Week 76 | -2.6 (13.8) | -1.7 (13.9)
  Week 84: number analyzed (Participants) | 148 | 35
  Week 84 | -3.4 (13.3) | -3.6 (13.8)
  Week 92: number analyzed (Participants) | 131 | 31
  Week 92 | -1.9 (13.2) | -1.8 (12.8)
  Week 100: number analyzed (Participants) | 125 | 29
  Week 100 | 0.0 (13.4) | 0.7 (12.0)
  Week 104: number analyzed (Participants) | 112 | 29
  Week 104 | -0.4 (12.6) | 0.0 (12.3)

47. Secondary Outcome: Change From BL to Each Study Visit in Serum HbA1c Level
Description: HbA1c was measured at each timepoint and presented in 'fraction of 1' unit by dividing the values in percentage by 100, in order to fit for CDISC (Clinical Data Interchange Standards Consortium) standard terminology. Changes from baseline to each timepoint were reported in unit 'fraction of 1'. Baseline was assessed on Day 1 visit. If baseline value was missing, the value from screening visit was used. In case of missing data, no imputation rules were applied.
Time Frame: Baseline and weeks 12, 28, 36, 44, 60, 84, 104
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Fraction of 1
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
Fraction of 1
  Week 12: number analyzed (Participants) | 338 | 182
  Week 12 | 0.0007 (0.0064) | -0.0001 (0.0061)
  Week 28: number analyzed (Participants) | 304 | 145
  Week 28 | 0.0006 (0.0086) | 0.0008 (0.0091)
  Week 36: number analyzed (Participants) | 225 | 108
  Week 36 | 0.0011 (0.0098) | 0.0007 (0.0075)
  Week 44: number analyzed (Participants) | 282 | 125
  Week 44 | 0.0018 (0.0081) | -0.0002 (0.0074)
  Week 60: number analyzed (Participants) | 200 | 70
  Week 60 | 0.0009 (0.0073) | 0.0012 (0.0080)
  Week 84: number analyzed (Participants) | 147 | 38
  Week 84 | 0.0028 (0.0085) | 0.0022 (0.0111)
  Week 104: number analyzed (Participants) | 111 | 29
  Week 104 | 0.0014 (0.0073) | 0.0004 (0.0059)

48. Secondary Outcome: Change From BL to Each Study Visit in Fasting Blood Glucose
Description: as for outcome 44
Time Frame: Baseline and weeks 4, 8, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 104
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 323 | 163
mmol/L
  Week 4: number analyzed (Participants) | 241 | 134
  Week 4 | 0.107 (2.573) | -0.076 (2.730)
  Week 8: number analyzed (Participants) | 233 | 128
  Week 8 | -0.103 (3.179) | -0.162 (3.118)
  Week 12: number analyzed (Participants) | 223 | 118
  Week 12 | -0.100 (3.504) | -0.153 (4.629)
  Week 20: number analyzed (Participants) | 211 | 99
  Week 20 | -0.302 (4.052) | 0.523 (2.981)
  Week 28: number analyzed (Participants) | 199 | 95
  Week 28 | 0.160 (3.489) | 0.045 (3.281)
  Week 36: number analyzed (Participants) | 185 | 83
  Week 36 | 0.015 (2.991) | -0.117 (2.812)
  Week 44: number analyzed (Participants) | 167 | 76
  Week 44 | 0.073 (2.683) | 0.801 (3.416)
  Week 52: number analyzed (Participants) | 168 | 79
  Week 52 | 0.048 (4.348) | -0.086 (4.883)
  Week 60: number analyzed (Participants) | 116 | 47
  Week 60 | 0.130 (2.907) | 1.190 (3.946)
  Week 68: number analyzed (Participants) | 91 | 33
  Week 68 | 0.185 (2.831) | 0.698 (3.386)
  Week 76: number analyzed (Participants) | 81 | 28
  Week 76 | -0.015 (2.031) | -0.671 (5.148)
  Week 84: number analyzed (Participants) | 75 | 20
  Week 84 | 0.495 (3.117) | 0.435 (2.037)
  Week 92: number analyzed (Participants) | 65 | 19
  Week 92 | 0.612 (2.494) | -0.861 (3.298)
  Week 100: number analyzed (Participants) | 58 | 19
  Week 100 | 0.405 (2.932) | -0.699 (2.161)
  Week 104: number analyzed (Participants) | 59 | 20
  Week 104 | 0.125 (2.633) | 0.237 (3.938)

49. Secondary Outcome: Change From BL to Each Study Visit in Albumin/Creatinine Ratio in Urine
Description: Baseline assessment was the assessment from day 1 visit. If baseline value was missing, value from screening visit was used. In case of missing data, no imputation rules were applied. To compute the geometric mean of albumin/creatinine ratio in urine and associated 95% CI, the mean of log-transformed albumin/creatinine ratio in urine values (ratio) and associated 95% CI are back-transformed to the raw scale. All assessments collected after initiation of dialysis (acute or chronic) were excluded from the analysis.
Time Frame: Baseline and weeks 12, 24, 36, 52, 64, 76, 88, 104
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 159 | 94
Ratio
  Week 12: number analyzed (Participants) | 122 | 75
  Week 12 | 1.08 [0.96 to 1.20] | 1.06 [0.84 to 1.34]
  Week 24: number analyzed (Participants) | 103 | 53
  Week 24 | 1.19 [1.04 to 1.36] | 1.16 [0.89 to 1.53]
  Week 36: number analyzed (Participants) | 90 | 49
  Week 36 | 1.21 [1.04 to 1.41] | 1.04 [0.77 to 1.40]
  Week 52: number analyzed (Participants) | 74 | 38
  Week 52 | 1.28 [1.02 to 1.59] | 1.04 [0.72 to 1.51]
  Week 64: number analyzed (Participants) | 22 | 11
  Week 64 | 1.25 [0.84 to 1.87] | 0.96 [0.53 to 1.71]
  Week 76: number analyzed (Participants) | 14 | 10
  Week 76 | 1.12 [0.51 to 2.44] | 0.82 [0.41 to 1.65]
  Week 88: number analyzed (Participants) | 11 | 2
  Week 88 | 1.10 [0.38 to 3.17] | 0.51 [0.27 to 0.97]
  Week 104: number analyzed (Participants) | 4 | 2
  Week 104 | 1.92 [0.75 to 4.89] | 0.38 [0.08 to 1.88]

50. Secondary Outcome: Change From BL to Each Study Visit in Serum Creatinine (Cr) Ratio
Description: Baseline assessment was the assessment from day 1 visit. If baseline value was missing, the value from screening visit was used. In case of missing data, no imputation rules were applied. To compute the geometric mean of serum Cr (ratio) and associated 95% CI, the mean of log-transformed serum Cr (ratio) values and associated 95% CI are back-transformed to the raw scale. All assessments collected after initiation of dialysis (acute or chronic) were excluded from the analysis.
Time Frame: Baseline and weeks 4, 8, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 104
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
Ratio
  Week 4: number analyzed (Participants) | 355 | 188
  Week 4 | 1.01 [1.00 to 1.03] | 1.05 [1.03 to 1.07]
  Week 8: number analyzed (Participants) | 338 | 184
  Week 8 | 1.03 [1.01 to 1.05] | 1.07 [1.04 to 1.09]
  Week 12: number analyzed (Participants) | 323 | 169
  Week 12 | 1.04 [1.02 to 1.06] | 1.07 [1.04 to 1.11]
  Week 20: number analyzed (Participants) | 289 | 135
  Week 20 | 1.08 [1.06 to 1.12] | 1.09 [1.05 to 1.13]
  Week 28: number analyzed (Participants) | 267 | 124
  Week 28 | 1.12 [1.08 to 1.16] | 1.13 [1.08 to 1.17]
  Week 36: number analyzed (Participants) | 238 | 108
  Week 36 | 1.12 [1.08 to 1.16] | 1.12 [1.07 to 1.18]
  Week 44: number analyzed (Participants) | 216 | 99
  Week 44 | 1.12 [1.07 to 1.16] | 1.16 [1.10 to 1.22]
  Week 52: number analyzed (Participants) | 201 | 90
  Week 52 | 1.12 [1.07 to 1.16] | 1.15 [1.09 to 1.22]
  Week 60: number analyzed (Participants) | 135 | 52
  Week 60 | 1.09 [1.05 to 1.14] | 1.15 [1.07 to 1.23]
  Week 68: number analyzed (Participants) | 117 | 36
  Week 68 | 1.11 [1.06 to 1.17] | 1.24 [1.13 to 1.37]
  Week 76: number analyzed (Participants) | 102 | 33
  Week 76 | 1.13 [1.07 to 1.20] | 1.23 [1.12 to 1.36]
  Week 84: number analyzed (Participants) | 94 | 26
  Week 84 | 1.13 [1.07 to 1.20] | 1.19 [1.05 to 1.35]
  Week 92: number analyzed (Participants) | 83 | 24
  Week 92 | 1.19 [1.12 to 1.27] | 1.22 [1.05 to 1.41]
  Week 100: number analyzed (Participants) | 75 | 22
  Week 100 | 1.16 [1.08 to 1.24] | 1.26 [1.06 to 1.50]
  Week 104: number analyzed (Participants) | 66 | 23
  Week 104 | 1.16 [1.05 to 1.27] | 1.28 [1.09 to 1.51]

51. Secondary Outcome: Time to Doubling of Serum Creatinine or Chronic Dialysis or Renal Transplant Compared to Baseline
Description: The endpoint was defined as time to doubling serum creatinine or chronic dialysis or renal transplant what ever came first. Time to event was defined as (First event date - Analysis date of first dose intake + 1) / 365.25. First event date was defined as date of dialysis or date of renal transplant (whichever occurred first) and analysis date of first dose intake was defined as date of first study drug dose intake collected on day 1 visit. Data analysis was completed using Kaplan-Meier estimate for cumulative proportion. The data evaluated until the safety emergent period, which was defined as the evaluation period from analysis date of first drug intake up to 28 days after the analysis last dose, and results were presented for every 6 months up to 2 years.
Time Frame: Baseline and year 0.5, year 1, year 1.5 and year 2
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
Percentage of participants
  Years 0.5 | 17.4 [13.4 to 21.4] | 17.8 [12.3 to 23.4]
  Years 1 | 36.8 [31.6 to 42.1] | 35.4 [27.9 to 42.9]
  Years 1.5 | 47.3 [41.4 to 53.1] | 48.2 [38.6 to 57.8]
  Years 2 | 55.0 [48.5 to 61.4] | 54.7 [43.8 to 65.6]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Time to doubling of serum Creatinine. Hazard ratio was calculated using stratified Cox Proportional Hazards Regression stratifying on CV history and region and adjusting on Hb and eGFR at baseline as continuous covariates; Test type: Superiority; p = 0.973, Regression, Cox; Hazard Ratio (HR) = 0.995, 95% CI 2-sided [0.75 to 1.32]

52. Secondary Outcome: Time to CKD Progression (Composite of Doubling Serum Creatinine, Chronic Dialysis or Renal Transplant, and Death)
Description: CKD progression was defined as date of occurrence of chronic dialysis or date of renal transplant or doubled serum creatinine or date of death, whichever came first. The time to CKD progression was calculated (in years) as (First event date - Analysis date of first dose intake + 1) / 365.25. First event date was defined as first occurrence of serum creatinine being doubled compared with baseline, first occurrence of chronic dialysis or renal transplant, occurrence of participants who died (whichever occurred first). Analysis date of first dose intake was defined as date of first study drug dose intake collected on day 1 visit. Data analysis was completed using Kaplan-Meier estimate for cumulative proportion. The data evaluated until the safety emergent period, which was defined as the evaluation period from analysis date of first drug intake up to 28 days after the analysis last dose, and results were presented for every 6 months up to 2 years.
Time Frame: Baseline and year 0.5, year 1, year 1.5 and year 2
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
Percentage of participants
  Years 0.5 | 20.5 [16.3 to 24.7] | 20.0 [14.2 to 25.8]
  Years 1 | 40.3 [35.1 to 45.5] | 38.3 [30.7 to 45.8]
  Years 1.5 | 50.2 [44.5 to 55.9] | 50.5 [41.1 to 59.9]
  Years 2 | 58.9 [52.7 to 65.1] | 61.1 [50.5 to 71.7]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Time to CKD progression. Hazard ratio was calculated using stratified Cox Proportional Hazards Regression stratifying on CV history and region and adjusting on Hb and eGFR at baseline as continuous covariates; Test type: Superiority; p = 0.972, Regression, Cox; Hazard Ratio (HR) = 0.995, 95% CI 2-sided [0.76 to 1.30]

53. Secondary Outcome: Time to at Least 40% Decrease in eGFR From Baseline, Chronic Dialysis or Renal Transplant
Description: All eGFR values collected during the safety emergent period are considered, excluding those collected on or after initiation of dialysis (acute or chronic). The First event date was defined as First occurrence of 40% decrease in eGFR from baseline, first occurrence of chronic dialysis or renal transplant (whichever occurred first and Analysis date of first dose intake was defined as date of first study drug dose intake collected on day 1 visit. The safety emergent period was defined as the evaluation period from the analysis date of first drug intake up to 28 days after the analysis date of last dose or end of study (EOS), whichever occurred first. Data analysis was completed using Kaplan-Meier estimate for cumulative proportion. The data evaluated until the safety emergent period, which was defined as the evaluation period from analysis date of first drug intake up to 28 days after the analysis last dose, and results were presented for every 6 months up to 2 years.
Time Frame: Baseline and year 0.5, year 1, year 1.5 and year 2
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 389 | 203
Percentage of participants
  Years 0.5 | 20.7 [16.5 to 25.0] | 22.3 [16.2 to 28.4]
  Years 1 | 44.4 [39.0 to 49.8] | 44.0 [36.2 to 51.7]
  Years 1.5 | 54.6 [48.9 to 60.4] | 62.8 [53.2 to 72.5]
  Years 2 | 64.5 [64.5 to 70.7] | 67.0 [56.8 to 77.1]
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.439, Regression, Cox; Hazard Ratio (HR) = 0.905, 95% CI 2-sided [0.70 to 1.16]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 28 days after the last dose of study drug (up to 108 weeks), and up to 2.836 years at maximum for all-cause mortality
Description: The safety emergent period was defined as the evaluation period from analysis date of first drug intake up to 28 days after the analysis last dose. All-cause mortality was monitored at any time after first administration of study drug to the end of the post-study follow-up, which includes deaths reported after the 28-day follow-up after the last dose of study drug.
Arm/Group | Roxadustat | Placebo
All-Cause Mortality (participants affected / at risk) | 45/391 | 20/203
Serious Adverse Events (participants affected / at risk) | 241/391 | 115/203
Other Adverse Events (participants affected / at risk) | 204/391 | 103/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roxadustat (N=391) | Placebo (N=203)
Anaemia (Blood and lymphatic system disorders) | 8 (10) | 7 (9)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 6 (6) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 3 (3)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 3 (3) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (4) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 3 (3) | 3 (4)
Cardiac failure congestive (Cardiac disorders) | 1 (2) | 1 (2)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 8 (8) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (4)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1) | 0 (0)
Hyperparathyroidism secondary (Endocrine disorders) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Asthenia (General disorders) | 1 (1) | 2 (2)
Catheter site haemorrhage (General disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 1 (1) | 1 (1)
Death (General disorders) | 4 (4) | 3 (3)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 2 (2)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Hepatic mass (Hepatobiliary disorders) | 1 (1) | 0 (0)
Steatohepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bursitis infective (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 4 (5) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 3 (3) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 2 (3) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Hepatic echinococciasis (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Meningoencephalitis herpetic (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (2) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 5 (6) | 1 (1)
Pneumonia (Infections and infestations) | 17 (21) | 12 (14)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis chronic (Infections and infestations) | 5 (5) | 2 (2)
Pyonephrosis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 6 (6) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 1 (1)
Vulvovaginitis (Infections and infestations) | 1 (1) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 14 (17) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fat embolism (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 21 (23) | 11 (15)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hypervolaemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to the mediastinum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 5 (5) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 4 (4) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenic syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 1 (1)
Vascular encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Device dislocation (Product Issues) | 1 (2) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (2) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (3)
Acute prerenal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Azotaemia (Renal and urinary disorders) | 10 (11) | 8 (10)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 135 (135) | 62 (63)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Eczema nummular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Leg amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 2 (2) | 1 (1)
Blood pressure inadequately controlled (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 0 (0)
Diabetic vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 1 (2)
Hypertensive crisis (Vascular disorders) | 4 (4) | 5 (5)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 2 (2) | 0 (0)
Thrombophlebitis (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roxadustat (N=391) | Placebo (N=203)
Anaemia (Blood and lymphatic system disorders) | 16 (17) | 31 (45)
Diarrhoea (Gastrointestinal disorders) | 32 (38) | 6 (9)
Nausea (Gastrointestinal disorders) | 34 (44) | 6 (6)
Asthenia (General disorders) | 18 (22) | 11 (13)
Oedema peripheral (General disorders) | 44 (53) | 21 (22)
Viral upper respiratory tract infection (Infections and infestations) | 38 (50) | 9 (15)
Glomerular filtration rate decreased (Investigations) | 24 (25) | 13 (13)
Hyperkalaemia (Metabolism and nutrition disorders) | 36 (48) | 13 (19)
Hyperuricaemia (Metabolism and nutrition disorders) | 9 (9) | 11 (11)
Iron deficiency (Metabolism and nutrition disorders) | 26 (26) | 8 (10)
Headache (Nervous system disorders) | 20 (21) | 10 (11)
Hypertension (Vascular disorders) | 85 (138) | 27 (44)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2016-06-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT01887600/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/00/NCT01887600/SAP_001.pdf